CLINICAL TRIAL: NCT07407959
Title: Clinical Evidence Generation of AI Enabled Fast, Accurate and Precise Screening and Staging of Benign vs Malignant Pelvic Abnormalities
Brief Title: Screening and Staging of Benign vs Malignant Pelvic Abnormalities
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MCBookwalter; NCI-2025-09210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-011490 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants undergo MRI on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study evaluates whether newly developed non-FDA approved image processing techniques [Adaptive Image Reconstruction (AIR Recon) Deep Learning (DL) and Sonic DL] can provide improved quality and decreased time compared to current scanning techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18
* For prostate group, any patient referred for prostate MR for screening purposes with no prior prostate related treatment or prior biopsy
* For endometriosis group, any patient referred for possible endometriosis evaluation (pre-surgical)

Exclusion Criteria:

* Individuals unable to undergo MRI imaging (MR-conditional or MR-nonconditional devices which would need additional procedures/conditions for scanning, pregnant people, individuals with implanted metal, etc.)
* Patient under the age of 18
* Patient who is unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, patients referred for prostate MR and patients referred for endometriosis evaluation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in image quality (healthy volunteers) | Baseline
  Three expert radiologists will read scans (blinded to technique) and provide qualitative feedback to score image quality for standard of care (SOC) imaging, SOC with AirRecon DL, SOC with Sonic DL, and SOC with AirRecon DL and Sonic DL. Reader scoring will use a 1-5 Likert scale (1-5; 1:poor, 5:excellent).
Improvement in scan time | Baseline
  Will be considered improved if the duration of the added imaging does not exceed 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Candice A. Bookwalter, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials